CLINICAL TRIAL: NCT04075149
Title: Does Treatment of Androgen Excess Using Spironolactone Improve Ovulatory Rates in Girls With Androgen Excess?
Acronym: CBS009
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: The Waterloo Foundation (Other)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Associate Professor of Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21768
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Polycystic Ovary Syndrome; Puberty Disorders; Ovulation Disorder
Keywords: PCOS; Polycystic Ovary Syndrome; ovulation; puberty; hyperandrogenemia; androgen excess
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: non-randomized cross-sectional, before and after intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spironolactone (Experimental): 16 weeks without medication, then 16 weeks with medication, then 12 months without medication; spironolactone 50 mg tablets: 50-100 mg orally twice daily (1.7-3.3 mg/kg/24 hr)
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — Spironolactone is an androgen-receptor commonly used (off-label) for hyperandrogenism in girls and women. It is used in this study to determine if androgen blockade can improve ovulation rates in girls with androgen excess, who often have low rates of ovulation in the years following menarche. The spironolactone dose will be as follows: If ≤ 60 kg, 50 mg twice daily; if > 60 kg, 100 mg twice daily.
  Other Names: Aldactone

SUMMARY:
Adolescent girls with androgen excess have a higher rate of irregular periods and decreased ovulation rates compared to normal girls, and are considered at-risk for developing polycystic ovary syndrome (PCOS). This pilot study will look at whether giving spironolactone might improve ovulation rates in girls with androgen excess, ages 13-19. If this is true, spironolactone treatment to young girls might prevent PCOS from developing and avoid future infertility.

DETAILED DESCRIPTION:
This is a non-randomized, clinical pilot study testing whether 16 weeks of spironolactone improves ovulation rates in post-menarcheal girls with androgen excess. The investigators will recruit girls ages 13-19 with clinical or biochemical androgen excess (defined as hirsutism and/or elevated Tanner stage-specific free testosterone concentrations) who are 4 to 6 years post-menarche. Girls will keep a menstrual diary and collect twice weekly saliva samples for progesterone and estradiol for 16 weeks before and for 16 weeks during spironolactone (if ≤ 60 kg, 50 mg twice daily; if > 60 kg, 100 mg twice daily [1.7-3.3 mg/kg/24 hr]) use. Girls will be asked to continue to collect saliva twice weekly for progesterone and estradiol testing for an additional 16 weeks after discontinuation of spironolactone and to continue menstrual diaries off of study medication for 12 additional months to assess persistence of any spironolactone effect. Ovulation events will be counted per 100 days based on definitive rises in salivary progesterone. The primary outcome will be changes in ovulation rate during spironolactone use compared to baseline. Changes in menstrual regularity via inter-menstrual interval will also be assessed as a secondary outcome of spironolactone administration. Another secondary outcome will be changes in acne and/or hirsutism.

ELIGIBILITY:
Inclusion Criteria:

* Girls age 13 - 19 years, with clinical or biochemical HA (defined as hirsutism and/or elevated Tanner stage-specific free testosterone concentrations) that are 4-6 years post-menarche
* Screening labs within age-appropriate normal range
* Volunteers who are 18-19 y old must be willing and able to provide written informed consent.
* When the subject is a minor (i.e., age < 18 y), the subject and custodial parents must be willing and able to provide written informed assent and consent, respectively.
* Willingness to strictly avoid pregnancy (using non-hormonal methods) during the time of study.

Exclusion Criteria:

* Age < 13 or > 19 y
* Girls ≤ 3 years and ≥ 7 years post-menarche will be excluded
* Being a study of androgen excess in adolescent girls with HA, men and boys are excluded
* Inability to comprehend what will be done during the study or why it will be done
* Precocious puberty (breast development before age 7)
* Primary amenorrhea (no menses by age 16)
* BMI-for-age < 5th percentile
* Patients currently enrolled in another research protocol will be excluded, except for those enrolled in IRB-HSR 17633 DENND1A
* Obesity due to genetic syndrome (e.g. Prader-Willi syndrome)
* Cushing syndrome
* Positive pregnancy test or lactation. Subjects with a positive pregnancy test will be informed of the result by the screening physician. Under Virginia law, parental notification is not required for minors. However, the screening physician will encourage them to tell their parent(s) and counsel them about the importance of appropriate prenatal care and counseling. We will arrange follow-up for them at the Teen Health Clinic at the University of Virginia or their primary care physician's office in a timely manner.
* Diabetes mellitus
* History of congenital adrenal hyperplasia or 17-hydroxyprogesterone > 300 ng/dL in the follicular phase, which suggests the possibility of congenital adrenal hyperplasia. NOTE: If a 17-hydroxyprogesterone > 300 ng/dL is confirmed on repeat testing, and ACTH-stimulated 17-hydroxyprogesterone < 1000 ng/dL will be required for study participation.
* Total testosterone > 150 ng/dL
* Abnormal thyroid stimulating hormone (TSH) for age. Subjects with adequately treated hypothyroidism, reflected by normal TSH values, will not be excluded.
* Abnormal sodium, potassium, or bicarbonate concentrations, or elevated creatine concentration (confirmed on repeat)
* Subjects must not take exogenous steroids or any medications known to affect the reproductive axis or glucose metabolism for 3 months prior to the study (or in the 2 months prior to screening). Such medications include oral contraceptives, progestins, metformin, glucocorticoids, and antipsychotic medications
* If sexually active, subjects will be required to abstain and/or use barrier forms of contraception during the study.

Note: Abnormal laboratory studies may be confirmed by repeat testing to exclude laboratory error.

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Ovulation Rate Changes | Rates of ovulation during weeks 17-32 (on medication) and weeks 33-48 (after medication) compared to weeks 1-16 (baseline, prior to medication)
  Ovulation rate during and after spironolactone compared to before medication. Ovulation will be counted based on salivary progesterone levels. The rate of ovulation will be defined as the number of ovulatory cycles per 100 days of follow-up.

SECONDARY OUTCOMES:
Menstrual Regularity Changes | IMI for weeks 1-16 (before medication, baseline), weeks 17-32 (on medication), and weeks 33-52 (after medication)
  Menstrual length during and after spironolactone compared to before medication. Changes in menstrual regularity will be assessed using inter-menstrual interval (IMI)
Acne | weeks 16 and 32
  Changes in acne before vs. after spironolactone treatment assessed using the Global Acne Grading System
Hirsutism | weeks 16 and 32
  Changes in hirsutism before vs. after spironolactone assessed using a modified Ferriman-Gallwey scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Christine Burt Solorzano, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Research in Reproduction, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No